CLINICAL TRIAL: NCT00556712
Title: A Randomized, Double-blind Study to Evaluate the Effect of Tarceva or Placebo Following Platinum-based CT on Overall Survival and Disease Progression in Patients With Advanced, Recurrent or Metastatic NSCLS Who Have Not Experienced Disease Progression or Unacceptable Toxicity During Chemotherapy
Brief Title: A Study of Tarceva (Erlotinib) Following Platinum-Based Chemotherapy in Patients With Advanced, Recurrent, or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BO18192
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Erlotinib (Experimental): Participants received erlotinib, 150 milligrams (mg), orally (PO), daily from randomization until progressive disease (PD), death, or unacceptable toxicity.
  Interventions: Drug: erlotinib [Tarceva]
- Placebo (Placebo Comparator): Participants received a placebo, PO, daily, from randomization until PD, death, or unacceptable toxicity.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: erlotinib [Tarceva] — 150mg po daily
  Arms: Erlotinib
Drug: Placebo — po daily
  Arms: Placebo

SUMMARY:
This 2 arm study will evaluate the efficacy, safety, and pharmacokinetics of Tarceva, compared with placebo, following platinum-based chemotherapy in patients with advanced, recurrent, or metastatic NSCLC who have not had disease progression or unacceptable toxicity during chemotherapy. Following 4 cycles of platinum-based chemotherapy, eligible patients will be randomized to receive either Tarceva 150mg po daily, or placebo daily. The anticipated time on study treatment is until disease progression; the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* histologically documented, locally advanced , recurrent or metastatic NSCLC;
* measurable disease;
* no disease progression after 4 cycles of platinum-based chemotherapy.

Exclusion Criteria:

* unstable systemic disease;
* any other malignancies in the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 889 (Actual)
Dates: Start 2006-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (113):
- Australia (8):
  - St Leonards, New South Wales
  - Waratah, New South Wales
  - Brisbane, Queensland
  - Adelaide, South Australia
  - East Bentleigh, Victoria
  - Fitzroy, Victoria
  - Geelong, Victoria
  - Melbourne, Victoria
- Austria (3):
  - Innsbruck
  - Klagenfurt
  - Vienna
- Belgium (2):
  - Antwerp
  - Edegem
- Canada (6):
  - Winnipeg, Manitoba
  - Oshawa, Ontario
  - Sault Ste. Marie, Ontario
  - Toronto, Ontario
  - Laval, Quebec
  - Montreal, Quebec
- Santiago, Chile
- China (3):
  - Beijing
  - Guangzhou
  - Shanghai
- Czechia (3):
  - České Budějovice
  - Olomouc
  - Pilsen
- Denmark (2):
  - Herlev
  - Odense
- France (11):
  - Bayonne
  - Brest
  - Clermont-Ferrand
  - Dijon
  - Le Mans
  - Lille
  - Limoges
  - Paris
  - Pau
  - Toulouse
  - Vandœuvre-lès-Nancy
- Germany (6):
  - Bad Berka
  - Bochum
  - Halle
  - Herne
  - Neuruppin
  - Villingen-Schwenningen
- Greece (2):
  - Athens
  - Heraklion
- Hungary (6):
  - Budapest
  - Deszk
  - Nyíregyháza
  - Pécs
  - Szombathely
  - Törökbálint
- Italy (3):
  - Bologna, Emilia-Romagna
  - Rome, Lazio
  - Ancona, The Marches
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Malaysia (2):
  - George Town
  - Kuala Lumpur
- Netherlands (4):
  - Amsterdam
  - Flushing
  - Heerlen
  - Nieuwegein
- New Zealand (2):
  - Auckland
  - Christchurch
- Poland (2):
  - Lodz
  - Otwock
- Romania (4):
  - Bucharest
  - Cluj-Napoca
  - Iași
  - Timișoara
- Russia (14):
  - Arkhangelsk
  - Balashikha
  - Chelyabinsk
  - Kazan'
  - Kirov
  - Krasnodar
  - Kuzmolovo
  - Moscow
  - Nizhny Novgorod
  - Perm
  - Saint Petersburg
  - Sashi
  - Smolensk
  - Yaroslavl
- Slovakia (4):
  - Banská Bystrica
  - Bratislava
  - Nitra
  - Poprad
- Slovenia (3):
  - Golnik
  - Ljubljana
  - Maribor
- South Africa (3):
  - Durban
  - Johannesburg
  - Pretoria
- South Korea (3):
  - Daegu
  - Seoul
  - Suwon
- Spain (5):
  - Santander, Cantabria
  - A Coruña, La Coruña
  - Oviedo, Principality of Asturias
  - Valencia, Valencia
  - Zaragoza, Zaragoza
- Ukraine (3):
  - Kharkiv
  - Uzhhorod
  - Zaporizhzhya
- United Kingdom (4):
  - Chelmsford
  - Dundee
  - Leicester
  - Plymouth
- Caracas, Venezuela

REFERENCES:
- [Derived] Cappuzzo F, Ciuleanu T, Stelmakh L, Cicenas S, Szczesna A, Juhasz E, Esteban E, Molinier O, Brugger W, Melezinek I, Klingelschmitt G, Klughammer B, Giaccone G; SATURN investigators. Erlotinib as maintenance treatment in advanced non-small-cell lung cancer: a multicentre, randomised, placebo-controlled phase 3 study. Lancet Oncol. 2010 Jun;11(6):521-9. doi: 10.1016/S1470-2045(10)70112-1. Epub 2010 May 20. PMID 20493771

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants completed 4 cycles (3 or 4 week cycles) of a standard platinum based non-investigational chemotherapy according to local practice and in concordance with the local labeling instructions (chemotherapy run-in period). Participants who completed all 4 cycles of chemotherapy run-in without progressive disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) were randomized to receive a placebo, orally (PO) as tablets, daily, from randomization until PD, death, unacceptable toxicity, or end of study, up to 27 months.
- Erlotinib, 150 Milligrams Per Day (mg/Day): Participants completed 4 cycles (3 or 4 week cycles) of a standard platinum based non-investigational chemotherapy according to local practice and in concordance with the local labeling instructions (chemotherapy run-in period). Participants who completed all 4 cycles of chemotherapy run-in without PD according to RECIST were randomized to receive erlotinib, 150 mg/day, PO as tablets from randomization until PD, death, unacceptable toxicity, or end of study, up to 27 months.
Period: Overall Study
Arm/Group | Placebo | Erlotinib, 150 Milligrams Per Day (mg/Day)
Started | 451 | 438
Completed | 0 (Data cutoff date: 17 May 2008) | 0 (Data cutoff date: 17 May 2008)
Not Completed | 451 | 438
Not completed — Adverse Event | 7 | 19
Not completed — Death | 5 | 10
Not completed — Progressive Disease | 383 | 320
Not completed — Protocol Violation | 3 | 2
Not completed — Refused Treatment | 17 | 16
Not completed — Failure to Return | 2 | 3
Not completed — Other | 2 | 2
Not completed — Ongoing at Data Cutoff | 32 | 66

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): all randomized participants presented according to the therapy that they were randomized to receive
Groups:
- Placebo: Participants completed 4 cycles (3 or 4 week cycles) of a standard platinum based non-investigational chemotherapy according to local practice and in concordance with the local labeling instructions (chemotherapy run-in period). Participants who completed all 4 cycles of chemotherapy run-in without PD according to RECIST were randomized to receive a placebo, PO as tablets, daily, from randomization until PD, death, unacceptable toxicity, or end of study, up to 27 months.
- Erlotinib, 150 mg/Day: Participants completed 4 cycles (3 or 4 week cycles) of a standard platinum based non-investigational chemotherapy according to local practice and in concordance with the local labeling instructions (chemotherapy run-in period). Participants who completed all 4 cycles of chemotherapy run-in without PD according to RECIST were randomized to receive erlotinib, 150 mg/day, PO as tablets from randomization until PD, death, unacceptable toxicity, or end of study, up to 27 months.
- Total: Total of all reporting groups
Arm/Group | Placebo | Erlotinib, 150 mg/Day | Total
Number analyzed (Participants) | 451 | 438 | 889
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (9.39) | 59.8 (9.52) | 59.8 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 117 | 230
  Male | 338 | 321 | 659

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With PD According to Response Evaluation Criteria in Solid Tumors (RECIST) or Death (Data Cutoff 17 May 2008)
Description: Progression-free survival (PFS) was defined as the time from randomization to PD or death, whichever occurred first. For target lesions (TLs), PD was defined at least a 20 percent (%) increase in the sum of the largest diameter (SLD), taking as reference the smallest SLD recorded from baseline (BL) more the appearance of one or more new lesions. For non-target lesions (NTLs), PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without PD or death were censored at the date of last tumor assessment where non-progression was documented.
Time Frame: Screening, BL [≤21 days after randomization], every 6 weeks thereafter until Week 48, every 12 weeks thereafter until PD, discontinuation of study treatment, or end of survival follow-up, up to data cutoff of 17 May 2008 (up to 27 months)
Population: FAS; participants with PD prior to randomization were excluded from analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 447 | 437
percentage of participants | 89.5 | 79.9

2. Primary Outcome: PFS in All Participants (Data Cutoff 17 May 2008)
Description: The median time, in weeks, from randomization to PFS event. Participants without PD or death were censored at the date of last tumor assessment where non-progression was documented. The 95% confidence interval (CI) was estimated using Kaplan-Meier methodology.
Time Frame: Screening, BL (≤21 days after randomization), every 6 weeks thereafter until Week 48, every 12 weeks thereafter until PD, discontinuation of study treatment, or end of survival follow-up, up to data cutoff of 17 May 2008 (up to 27 months)
Population: FAS; participants with PD prior to randomization were excluded from analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 447 | 437
weeks | 11.1 [8.1 to 11.7] | 12.3 [12.0 to 13.3]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib, 150 mg/Day; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.62 to 0.82]

3. Primary Outcome: Probable Percentage of Participants Remaining Alive and Free of Disease Progression at 6 Months (Data Cutoff 17 May 2008)
Description: PFS was defined as the time from randomization to PD or death, whichever occurred first. For TLs, PD was defined at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from BL more the appearance of one or more new lesions. For NTLs, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without PD or death were censored at the date of last tumor assessment where non-progression was documented. The 95% CI was estimated using Kaplan-Meier methodology.
Time Frame: 6 months
Population: FAS; participants with PD prior to randomization were excluded from analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 447 | 437
percentage of participants | 15.0 [12.0 to 19.0] | 25.0 [21.0 to 29.0]

4. Primary Outcome: Percentage of Epidermal Growth Factor Receptor (EGFR) Immunohistochemistry (IHC) Positive Participants With PD or Death (Data Cutoff 17 May 2008)
Description: PFS was defined as the time from randomization to PD or death, whichever occurred first. For TLs, PD was defined at least a 20% increase in the SLD, taking as reference the smallest SLD recorded since treatment started or the appearance of one or more new lesions. For NTLs, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without PD or death were censored at the date of last tumor assessment where non-progression was documented.
Time Frame: as for outcome 2
Population: FAS; only participants with EGFR IHC positive tumors were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 311 | 307
percentage of participants | 89.4 | 79.5

5. Secondary Outcome: Percentage of All Participants Who Died (Data Cutoff 12 January 2012)
Time Frame: Screening, BL (≤21 days after randomization), every 6 weeks thereafter until Week 48, every 12 weeks thereafter until PD, discontinuation of study treatment, or end of survival follow-up, up to data cutoff of 12 January 2012 (up to 71 months).
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 451 | 438
percentage of participants | 87.1 | 82.0

6. Secondary Outcome: Overall Survival (OS) in All Participants (Data Cutoff 12 January 2012)
Description: OS was defined as the median time, in months, from the date of randomization to the date of death, due to any cause. Patients who have not died at the time of the final analysis will be censored at the date the patient was last known to be alive. The 95% CI was estimated using Kaplan-Meier methodology.
Time Frame: Screening, BL (≤ 21 days after randomization), every 6 weeks thereafter until Week 48, every 12 weeks thereafter until PD, discontinuation of study treatment, or end of survival follow-up, up to data cutoff of 12 January 2012 (up to 71 months)
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 451 | 438
months | 11.0 [9.9 to 12.0] | 12.4 [10.6 to 13.9]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib, 150 mg/Day; Test type: Superiority or Other; p = 0.0097, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.72 to 0.96]

7. Secondary Outcome: Probable Percentage of Participants Remaining Alive at 1 Year (Data Cutoff 12 January 2012)
Description: as for outcome 6
Time Frame: 1 year
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 451 | 438
percentage of participants | 45.0 [41.0 to 50.0] | 50.0 [45.0 to 55.0]

8. Secondary Outcome: Percentage of EGFR IHC Positive Participants Who Died (Data Cutoff 12 January 2012)
Time Frame: as for outcome 5
Population: FAS; only participants with EGFR IHC positive tumors were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 313 | 308
percentage of participants | 87.5 | 80.5

9. Secondary Outcome: OS in EGFR IHC Positive Population (Data Cutoff 12 January 2012)
Description: as for outcome 6
Time Frame: as for outcome 5
Population: FAS; only participants with EGFR IHC positive tumors were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 313 | 308
months | 11.0 [9.7 to 12.8] | 12.8 [11.1 to 14.7]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib, 150 mg/Day; Test type: Superiority or Other; p = 0.0050, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.66 to 0.93]

10. Secondary Outcome: Probable Percentage of Participants in the EGFR IHC Positive Population Remaining Alive at 1 Year (Data Cutoff 12 January 2012)
Description: as for outcome 6
Time Frame: 1 year
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 313 | 308
percentage of participants | 47.0 [41.0 to 52.0] | 52.0 [47.0 to 58.0]

11. Secondary Outcome: Percentage of EGFR IHC Negative Participants With PD or Death (Data Cutoff 17 May 2008)
Description: as for outcome 4
Time Frame: Screening, BL (≤21 days after randomization), every 6 weeks thereafter until Week 48, every 12 weeks thereafter until PD, discontinuation of study treatment, or end of survival follow-up, up to data cutoff of 17 May 2008 (up to 71 months)
Population: FAS; only participants with EGFR IHC negative tumors were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 59 | 62
percentage of participants | 89.8 | 77.4

12. Secondary Outcome: PFS in EGFR IHC Negative Participants (Data Cutoff 17 May 2008)
Description: The median time, in weeks, from randomization to PFS event. Participants without PD or death were censored at the date of last tumor assessment where non-progression was documented. The 95% CI was estimated using Kaplan-Meier methodology.
Time Frame: as for outcome 2
Population: FAS; only participants with EGFR IHC negative tumors were included in the analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 59 | 62
weeks | 9.0 [6.4 to 12.0] | 11.0 [6.6 to 13.1]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib, 150 mg/Day; Test type: Superiority or Other; p = 0.1768, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.51 to 1.14]

13. Secondary Outcome: Probable Percentage of Participants in the EGFR IHC Negative Population Remaining Alive and Free of Disease Progression at 6 Months (Data Cutoff 17 May 2008)
Description: PFS was defined as the time from randomization to PD or death, whichever occurred first. For TLs, PD was defined at least a 20% increase in the SLD, taking as reference the smallest SLD recorded since treatment started or the appearance of one or more new lesions. For NTLs, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without PD or death were censored at the date of last tumor assessment where non-progression was documented. The 95% CI was estimated using Kaplan-Meier methodology.
Time Frame: 6 months
Population: FAS; only participants with EGFR IHC negative tumors were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 59 | 62
percentage of participants | 11.0 [2.0 to 20.0] | 22.0 [11.0 to 34.0]

14. Secondary Outcome: Percentage of EGFR IHC Negative Participants Who Died (Data Cutoff 17 May 2008)
Time Frame: as for outcome 2
Population: FAS; only participants with EGFR IHC negative tumors were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 59 | 62
percentage of participants | 50.8 | 41.9

15. Secondary Outcome: OS in EGFR IHC Negative Participants (Data Cutoff 17 May 2008)
Description: as for outcome 6
Time Frame: as for outcome 2
Population: FAS; only participants with EGFR IHC negative tumors were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 59 | 62
months | 10.2 [7.4 to 11.2] | 8.6 [7.4 to NA] — The upper limit of the 95% CI could not be calculated due to the large number of censored events.
Statistical Analysis 1: Comparison: Placebo vs Erlotinib, 150 mg/Day; Test type: Superiority or Other; p = 0.4797, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.49 to 1.40]

16. Secondary Outcome: Probable Percentage of Participants in the EGFR IHC Negative Population Remaining Alive at 1 Year (Data Cutoff 17 May 2008)
Description: as for outcome 6
Time Frame: 1 year
Population: FAS; only participants with EGFR IHC negative tumors were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 59 | 62
percentage of participants | 20.0 [3.0 to 37.0] | 42.0 [25.0 to 59.0]

17. Secondary Outcome: Time to Progression (Data Cutoff 17 May 2008)
Description: The median time, in weeks, between randomization and TTP event. Participants without PD were censored at the date of last tumor assessment where non-progression was documented. If a participant received a second anti-cancer therapy without prior documentation of PD, the participant was censored at the date of last tumor assessment before starting new chemotherapy.
Time Frame: as for outcome 2
Population: FAS; participants with PD prior to randomization were excluded from analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 447 | 437
weeks | 11.3 [8.1 to 11.9] | 12.3 [12.0 to 14.1]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib, 150 mg/Day; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.61 to 0.82]

18. Secondary Outcome: Probable Percentage of Participants Remaining Progression-Free in the TTP Analysis at 6 Months (Data Cutoff 17 May 2008)
Description: TTP was defined as the time from the date of randomization to the first date PD was recorded. For TLs, PD was defined at least a 20% increase in the SLD, taking as reference the smallest SLD recorded since treatment started or the appearance of one or more new lesions. For NTLs, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without PD were censored at the date of last tumor assessment where non-progression was documented. If a participant received a second anti-cancer therapy without prior documentation of PD, the participant was censored at the date of last tumor assessment before starting new chemotherapy. The 95% CI was estimated using Kaplan-Meier methodology.
Time Frame: 6 months
Population: FAS; participants with PD prior to randomization were excluded from analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 447 | 437
percentage of participants | 15.0 [11.0 to 19.0] | 26.0 [21.0 to 30.0]

19. Secondary Outcome: Percentage of Participants With a Best Overall Response (BOR) of Confirmed Complete Response (CR) or Partial Response (PR) According to RECIST (Data Cutoff 17 May 2008)
Description: BOR was defined as CR or PR confirmed by repeat assessments performed no less than 4 weeks after the criteria for response was first met. For TLs, CR was defined as the disappearance of all TLs, and PR was defined as at least a 30% decrease in the SLD of the TLs, taking as a reference the baseline (BL) SLD. For NTLs, CR was defined as the disappearance of all NTLs and normalization of tumor marker levels. The 95% CI for one sample binomial was determined using the Pearson-Clopper method.
Time Frame: as for outcome 2
Population: FAS; only participants with CR, PR or SD at BL as determined by the Investigator were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 445 | 436
percentage of participants | 5.4 [3.5 to 7.9] | 11.9 [9.0 to 15.3]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib, 150 mg/Day; Test type: Superiority or Other; p = 0.0006, Chi-squared; Difference in Response Rates = 6.53, 95% CI 2-sided [2.7 to 10.3] — The approximate 95% CI for the difference of two rates was determined using the Hauck-Anderson method

20. Secondary Outcome: Percentage of Participants With a CR, PR, Stable Disease (SD), or PD According to RECIST (Data Cutoff 17 May 2008)
Description: For TLs, CR was defined as the disappearance of all TLs; PR was defined as at least a 30% decrease in the SLD of the TLs, taking as a reference the BL SLD; SD was defined as neither sufficient decrease in SLD to qualify for PR nor sufficient increase in SLD to qualify for PD; and PD was defined as at least a 20% increase in the SLD of TLs, taking as reference the smallest SLD recorded since the treatment started. For NTLs, CR was defined as the disappearance of all NTLs and normalization of tumor marker levels; SD/incomplete response was defined as the persistence of 1 or more NTLs and/or maintenance of tumor marker levels above normal limits; and PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. The 95% CI for one sample binomial was determined using the Pearson-Clopper method.
Time Frame: as for outcome 2
Population: FAS; only participants with CR, PR or SD at BL as determined by the Investigator were included in the analysis; and 7 and 17 participants were not assessed from the Placebo and Erlotinib, 150 mg/day groups, respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 445 | 436
percentage of participants
  CR | 0.7 [0.1 to 2.0] | 0.9 [0.3 to 2.3]
  PR | 4.7 [2.9 to 7.1] | 11.0 [8.2 to 14.3]
  SD | 45.4 [40.7 to 50.1] | 48.6 [43.8 to 53.4]
  PD | 47.6 [42.9 to 52.4] | 35.6 [31.1 to 40.2]

21. Secondary Outcome: Percentage of Participants With a Response Upgrade From BL According to RECIST (Data Cutoff 17 May 2008)
Description: Response upgrade was defined by a change of PR to CR or of SD to PR or CR from BL to the end of treatment. For TLs, CR was defined as the disappearance of all TLs; PR was defined as at least a 30% decrease in the SLD of the TLs, taking as a reference the BL SLD; SD was defined as neither sufficient decrease in SLD to qualify for PR nor sufficient increase in SLD to qualify for PD; and PD was defined as at least a 20% increase in the SLD of TLs, taking as reference the smallest SLD recorded since the treatment started. For NTLs, CR was defined as the disappearance of all NTLs and normalization of tumor marker levels; SD/incomplete response was defined as the persistence of 1 or more NTLs and/or maintenance of tumor marker levels above normal limits; and PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. The 95% CI for one sample binomial was determined using the Pearson-Clopper method.
Time Frame: as for outcome 2
Population: FAS; only participants with CR, PR or SD at BL as determined by the Investigator were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 445 | 436
percentage of participants | 1.3 [0.5 to 2.9] | 5.5 [3.6 to 8.1]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib, 150 mg/Day; Test type: Superiority or Other; p = 0.0007, Chi-squared; Difference in Response Upgrade Rates = 4.2, 95% CI 2-sided [1.6 to 6.7] — The approximate 95% CI for the difference of two rates was determined using the Hauck-Anderson method

22. Secondary Outcome: Percentage of Participants With a Change of PR to CR or SD to PR or CR From BL to End of Treatment According to RECIST (Data Cutoff 17 May 2008)
Description: as for outcome 20
Time Frame: as for outcome 2
Population: FAS; only participants with CR, PR or SD at BL as determined by the Investigator were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 445 | 436
percentage of participants
  PR to CR | 0.4 [0.1 to 1.6] | 0.5 [0.1 to 1.6]
  SD to PR | 0.9 [0.2 to 2.3] | 4.8 [3.0 to 7.3]
  SD to CR | 0.0 [0.0 to 0.8] | 0.2 [0.0 to 1.3]

23. Secondary Outcome: Percentage of Participants With CR, PR, or SD or With SD [Maintained For Greater Than (>) 12 Weeks] or CR or PR (Data Cutoff 17 May 2008)
Description: Disease control was defined as a best response of CR or PR or SD or a best response of SD for more than 12 weeks, or CR or PR. For TLs, CR was defined as the disappearance of all TLs; PR was defined as at least a 30% decrease in the SLD of the TLs, taking as a reference the BL SLD; SD was defined as neither sufficient decrease in SLD to qualify for PR nor sufficient increase in SLD to qualify for PD. For NTLs, CR was defined as the disappearance of all NTLs and normalization of tumor marker levels; SD/incomplete response was defined as the persistence of 1 or more NTLs and/or maintenance of tumor marker levels above normal limits. The 95% CI for one sample binomial was determined using the Pearson-Clopper method.
Time Frame: as for outcome 2
Population: FAS; only participants with CR, PR or SD at BL as determined by the Investigator were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 445 | 436
percentage of participants
  CR Plus (+) PR + SD | 50.8 [46.0 to 55.5] | 60.6 [55.8 to 65.2]
  CR + PR + SD >12 Weeks | 27.4 [23.3 to 31.8] | 40.8 [36.2 to 45.6]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib, 150 mg/Day; Analysis included CR + PR + SD rate; Test type: Superiority or Other; p = 0.0035, Chi-squared; Difference in Disease Control Rates = 9.8, 95% CI 2-sided [3.1 to 16.4] — Approximate 95% CI for the difference of two rates was determined using the Hauck-Anderson method
Statistical Analysis 2: Comparison: Placebo vs Erlotinib, 150 mg/Day; Analysis included CR + PR + SD > 12 weeks rate; Test type: Superiority or Other; p < 0.0001, Chi-squared; Difference in Disease Control Rates = 13.4, 95% CI 2-sided [7.1 to 19.7] — Approximate 95% CI for the difference of two rates was determined using the Hauck-Anderson method

24. Secondary Outcome: Percentage of Participants With Symptom Progression Assessed Using the Lung Cancer Subscale (LCS) (Data Cutoff 17 May 2008)
Description: LCS scores were obtained from a 7-item questionnaire from the Functional Assessment of Cancer Therapy - Lung (FACT-L) version (V) 4. Participants responded to questions assessing symptoms commonly reported by lung cancer patients; such as shortness of breath, loss of weight, and tightness in chest; on a scale from 0-4, where 0 equaled (=) "not at all" and 4 = "very much." The participants' responses were summed to result in an overall score, where a higher score indicated more severe symptoms. A change of 2 to 3 points in score was determined to be a clinically meaningful decline.
Time Frame: as for outcome 2
Population: FAS; 56 and 48 participants were not evaluated for this outcome measure from the Placebo and Erlotinib groups, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 395 | 390
percentage of participants | 44.1 | 47.7

25. Secondary Outcome: Time to Symptom Progression (Data Cutoff 17 May 2008)
Description: The median time, in weeks, from the date of randomization to the date of documented clinically meaningful decline in LCS from BL or death, whichever occurred first. LCS scores were obtained from a 7-item questionnaire from the FACT-L V 4. Participants responded to questions assessing symptoms commonly reported by lung cancer patients; such as shortness of breath, loss of weight, and tightness in chest; on a scale from 0-4, where 0 = "not at all" and 4 = "very much." The participants' responses were summed to result in an overall score, where a higher score indicated more severe symptoms. A change of 2 to 3 points in score was determined to be a clinically meaningful decline. The 95% CI was determined using Kaplan-Meier methodology.
Time Frame: as for outcome 2
Population: FAS
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 395 | 390
weeks | 17.6 [12.4 to 19.1] | 18.3 [13.1 to 24.1]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib, 150 mg/Day; Test type: Superiority or Other; p = 0.3787, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.74 to 1.12]

26. Secondary Outcome: Probable Percentage of Participants Remaining Without Symptom Progression at 6 Months (Data Cutoff 17 May 2008)
Description: LCS scores were obtained from a 7-item questionnaire from the FACT-L V 4. Participants responded to questions assessing symptoms commonly reported by lung cancer patients; such as shortness of breath, loss of weight, and tightness in chest; on a scale from 0-4, where 0 = "not at all" and 4 = "very much." The participants' responses were summed to result in an overall score, where a higher score indicated more severe symptoms. A change of 2 to 3 points in score was determined to be a clinically meaningful decline. The 95% CI was estimated using Kaplan-Meier methodology.
Time Frame: 6 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 395 | 390
percentage of participants | 35.0 [27.0 to 42.0] | 41.0 [34.0 to 47.0]

27. Primary Outcome: PFS in EGFR IHC Positive Population (Data Cutoff 17 May 2008)
Description: as for outcome 12
Time Frame: Screening, BL (≤ 21 days after randomization), every 6 weeks thereafter until Week 48, every 12 weeks thereafter until PD, discontinuation of study treatment, or end of survival follow-up, up to data cutoff of 17 May 2008 (up to 27 months)
Population: FAS;only participants with EGFR IHC positive tumors were included in the analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 311 | 307
weeks | 11.1 [7.1 to 11.7] | 12.3 [12.0 to 17.7]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib, 150 mg/Day; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.58 to 0.82]

28. Primary Outcome: Probable Percentage of Participants in the EGFR IHC Positive Population Remaining Alive and Progression Free at 6 Months (Data Cutoff 17 May 2008)
Description: as for outcome 13
Time Frame: 6 months
Population: FAS; only participants with EGFR IHC positive tumors were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 311 | 307
percentage of participants | 16.0 [12.0 to 21.0] | 27.0 [22.0 to 32.0]

29. Secondary Outcome: Percentage of Participants With Deterioration Assessed Using the Trial Outcome Index (Data Cutoff 17 May 2008)
Description: The Trial Outcome Index (TOI) was defined as the sum of the scores of the Physical Well-Being (PWB), Functional Well-Being (FWB), and LCS. PWB, FWB, and LCS scores were obtained from 7-item questionnaires from the FACT-L V 4. Participants responded to questions assessing symptoms on a scale from 0-4, where 0 = "not at all" and 4 = "very much." Higher score indicated more severe symptoms. A clinically meaningful decline in TOI score was defined as at least a 6 point decline from BL. Participants without a clinically meaningful decline in TOI at the time of analysis were censored at the time of the last FACT-L assessment.
Time Frame: as for outcome 2
Population: FAS; 59 and 49 participants were not evaluated for this outcome measure from the Placebo and Erlotinib groups, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 392 | 389
percentage of participants | 43.1 | 50.9

30. Secondary Outcome: Time to Deterioration in TOI (Data Cutoff 17 May 2008)
Description: The median time, in weeks, from the date of randomization until a clinically meaningful decline from BL in TOI or death, whichever occurred first. TOI was defined as the sum of PWB, FWB, and LCS scores, which were obtained from 7-item questionnaires from the FACT-L V 4. Participants responded to questions assessing symptoms on a scale from 0-4, where 0 = "not at all" and 4 = "very much." Higher score indicated more severe symptoms. A clinically meaningful decline in TOI score was defined as at least a 6 point decline from BL Participants without a clinically meaningful decline in TOI at the time of analysis were censored at the time of the last FACT-L assessment. The 95% CI was determined using Kaplan-Meier methodology.
Time Frame: as for outcome 2
Population: FAS
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 392 | 389
weeks | 18.9 [13.6 to 24.1] | 18.1 [12.3 to 19.0]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib, 150 mg/Day; Test type: Superiority or Other; p = 0.5385, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.87 to 1.31]

31. Secondary Outcome: Probable Percentage of Participants Remaining Without Deterioration in TOI at 6 Months (Data Cutoff 17 May 2008)
Description: TOI was defined as the sum of the scores of the PWB, FWB, and LCS. PWB, FWB, and LCS scores were obtained from 7-item questionnaires from the FACT-L V 4. Participants responded to questions assessing symptoms on a scale from 0-4, where 0 = "not at all" and 4 = "very much." Higher score indicated more severe symptoms. A clinically meaningful decline in TOI score was defined as at least a 6 point decline from BL. Participants without a clinically meaningful decline in TOI at the time of analysis were censored at the time of the last FACT-L assessment. The 95% CI was estimated using Kaplan-Meier methodology.
Time Frame: 6 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 392 | 389
percentage of participants | 41.0 [34.0 to 48.0] | 39.0 [33.0 to 45.0]

32. Secondary Outcome: Percentage of Participants With Deterioration in Quality of Life Assessed Using TOI, SWB, and EWB (Data Cutoff 17 May 2008)
Description: Deterioration in quality of life (QoL) was defined as a clinically meaningful decline in the total FACT-L score, the sum of the TOI, Social/Family Well-Being (SWB) and Emotional Well-Being (EWB) of the FACT-L questionnaires. TOI (PWB + FWB + LCS), SWB and EWB scores were obtained from 7-item (6-item in the case of EWB) questionnaires from the FACT-L V 4. Participants responded to questions assessing symptoms on a scale from 0-4, where 0 = "not at all" and 4 = "very much." Higher score indicated more severe symptoms. A clinically meaningful decline in FACT-L score was defined as at least a 6 point decline from BL. Participants without a clinically meaningful decline in TOI at the time of analysis were censored at the time of the last FACT-L.
Time Frame: as for outcome 2
Population: FAS; 62 and 51 participants were not evaluated for this outcome measure from the Placebo and Erlotinib groups, respectively,
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 389 | 387
percentage of participants | 51.7 | 55.3

33. Secondary Outcome: Time to Deterioration in QoL (Data Cutoff 17 May 2008)
Description: The median time, in weeks, from the date of randomization until a clinically meaningful decline from BL in total FACT-L or death, whichever occurred first. Total FACT-L score was defined as the sum of the TOI, SWB and EWB of the FACT-L questionnaires. TOI (PWB + FWB + LCS), SWB and EWB scores were obtained from 7-item (6-item in the case of EWB) questionnaires from the FACT-L V 4. Participants responded to questions assessing symptoms on a scale from 0-4, where 0 = "not at all" and 4 = "very much." Higher score indicated more severe symptoms. A clinically meaningful decline in FACT-L score was defined as at least a 6 point decline from BL. Participants without a clinically meaningful decline in TOI at the time of analysis were censored at the time of the last FACT-L assessment. The 95% CI was determined using Kaplan-Meier methodology.
Time Frame: as for outcome 2
Population: FAS
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 389 | 387
weeks | 12.3 [11.9 to 17.9] | 12.6 [12.1 to 18.1]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib, 150 mg/Day; Test type: Superiority or Other; p = 0.6530, Log Rank; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.79 to 1.16]

34. Secondary Outcome: Probable Percentage of Participants Remaining Without Deterioration in QoL at 6 Months (Data Cutoff 17 May 2008)
Description: Deterioration in QoL was defined as a clinically meaningful decline in the total FACT-L score, the sum of the TOI, SWB and EWB of the FACT-L questionnaires. TOI (PWB + FWB + LCS), SWB and EWB scores were obtained from 7-item (6-item in the case of EWB) questionnaires from the FACT-L V 4. Participants responded to questions assessing symptoms on a scale from 0-4, where 0 = "not at all" and 4 = "very much." Higher score indicated more severe symptoms. A clinically meaningful decline in FACT-L score was defined as at least a 6 point decline from BL. Participants without a clinically meaningful decline in TOI at the time of analysis were censored at the time of the last FACT-L. The 95% CI was estimated using Kaplan-Meier methodology.
Time Frame: 6 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 389 | 387
percentage of participants | 34.0 [27.0 to 40.0] | 32.0 [26.0 to 38.0]

35. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Lung (FACT-L) Scores (Data Cutoff 17 May 2008)
Description: Total FACT-L score=sum of TOI, SWB, and EWB of FACT-L questionnaires. TOI (PWB+FWB+LCS), SWB, and EWB scores obtained from 7-item (6-item for EWB) questionnaires from FACT-L V4. Participants responded to questions assessing symptoms (scale 0-4; 0="not at all" and 4="very much"). Higher score=more severe symptoms. The 7-item LCS assessed symptoms such as shortness of breath, loss of weight, tightness in chest. Participants responded to questions assessing symptoms (scale: 0-4; 0="not at all" and 4="very much"). Scores from 0-35; higher score=more severe symptoms. The 27 items of FACT-G were scored in the following domains: PWB (7 items, total score 0-28), SWB (7 items; total score 0-28), EWB (6 items, total score 0-24), and FWB (7 items; total score 0-28), higher scores=better QoL. Participants responded to items on 5-point Likert scale (0="Not at all" to 4="Very much"; total score: 0-108). Higher score=better QOL. TOI score=PWB+FWB+LCS; Total TOI score: 0-92; higher scores=better QOL.
Time Frame: as for outcome 2
Population: FAS; n=number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 397 | 392
score on a scale
  BL: Physical Well-Being (n=397,392) | 20.85 (4.817) | 20.96 (4.781)
  BL: Social Well-Being (n=397,392) | 20.84 (5.496) | 20.98 (5.285)
  BL: Emotional Well-Being (n=397,393) | 16.92 (4.534) | 16.77 (4.862)
  BL: Functional Well-Being (n=397,393) | 16.15 (5.488) | 16.84 (5.514)
  BL: FACT-L Subscale Score (n=397,391) | 24.17 (4.892) | 24.46 (4.697)
  BL: Lung Cancer Subscale Score (n=397,391) | 19.82 (4.188) | 20.07 (4.240)
  BL: Total FACT-General (FACT-G) Score (n=396,391) | 74.68 (14.787) | 75.52 (14.612)
  BL: Trial Outcome Index (n=396,390) | 56.83 (11.830) | 57.90 (11.682)
  BL: Total FACT-L Score (n=395,389) | 98.85 (18.007) | 100.02 (17.751)
  Week 6: Physical Well-Being (n=274,304) | 21.44 (5.117) | 20.69 (5.180)
  Week 6: Social Well-Being (n=274,303 | 20.62 (5.437) | 21.43 (5.178)
  Week 6: Emotional Well-Being (n=275,302) | 16.53 (4.587) | 17.17 (4.748)
  Week 6: Functional Well-Being (n=275,302) | 16.41 (5.234) | 16.87 (5.614)
  Week 6: FACT-L Subscale Score (n=275,300) | 24.45 (5.231) | 24.80 (5.000)
  Week 6: Lung Cancer Subscale Score (n=275,300) | 19.78 (4.463) | 20.13 (4.336)
  Week 6: Total FACT-G Score (n=274,300) | 74.82 (14.380) | 76.14 (15.132)
  Week 6: Trial Outcome Index (n=274,299) | 57.59 (12.292) | 57.64 (12.482)
  Week 6: Total FACT-L Score (n=274,297) | 99.27 (17.857) | 100.95 (18.360)
  Week 12: Physical Well-Being (n=144,194) | 21.93 (4.734) | 20.78 (5.368)
  Week 12: Social Well-Being (n=143,194) | 20.38 (5.637) | 20.04 (5.691)
  Week 12: Emotional Well-Being (n=144,194) | 17.21 (4.376) | 16.85 (4.521)
  Week 12: Functional Well-Being (n=144,196) | 17.04 (5.770) | 16.35 (5.745)
  Week 12: FACT-L Subscale Score (n=144,196) | 25.15 (4.735) | 24.19 (5.323)
  Week 12: Lung Cancer Subscale Score (n=144,196) | 20.22 (4.015) | 19.50 (4.600)
  Week 12: Total FACT-G Score (n=144,192) | 76.42 (14.889) | 74.06 (15.754)
  Week 12: Trial Outcome Index (n=144,194) | 59.19 (12.129) | 56.57 (13.276)
  Week 12: Total FACT-L Score (n=144,192) | 101.56 (17.824) | 98.30 (19.337)
  Week 18: Physical Well-Being (n=86,143) | 21.60 (4.883) | 21.40 (4.945)
  Week 18: Social Well-Being (n=86,143) | 21.08 (5.328) | 19.94 (6.130)
  Week 18: Emotional Well-Being (n=86,143) | 17.33 (4.717) | 17.14 (4.356)
  Week 18: Functional Well-Being (n=86,143) | 16.89 (5.289) | 16.83 (5.553)
  Week 18: FACT-L Subscale Score (n=86,143) | 25.44 (4.645) | 24.52 (5.344)
  Week 18: Lung Cancer Subscale Score (n=86,143) | 20.28 (4.003) | 19.64 (4.635)
  Week 18: Total FACT-G Score (n=86,143) | 76.89 (14.385) | 75.31 (16.648)
  Week 18: Trial Outcome Index (n=86,143) | 58.76 (11.492) | 57.87 (12.803)
  Week 18: Total FACT-L Score (n=86,143) | 102.33 (17.502) | 99.83 (20.558)
  Week 24: Physical Well-Being (n=59,101) | 21.78 (4.665) | 21.21 (4.898)
  Week 24: Social Well-Being (n=59,101) | 20.79 (5.641) | 20.49 (5.251)
  Week 24: Emotional Well-Being (n=59,100) | 16.86 (4.880) | 16.54 (4.615)
  Week 24: Functional Well-Being (n=59,100) | 17.14 (6.062) | 17.23 (5.300)
  Week 24: FACT-L Subscale Score (n=59,101) | 25.18 (5.126) | 25.13 (5.245)
  Week 24: Lung Cancer Subscale Score (n=59,101) | 20.07 (4.246) | 19.94 (4.487)
  Week 24: Total FACT-G Score (n=59,99) | 76.58 (16.091) | 75.50 (15.754)
  Week 24: Trial Outcome Index (n=59,100) | 58.99 (11.837) | 58.37 (12.686)
  Week 24: Total FACT-L Score (n=59,99) | 101.75 (19.347) | 100.69 (19.831)
  Week 30: Physical Well-Being (n=37,66) | 21.74 (4.153) | 21.77 (4.576)
  Week 30: Social Well-Being (n=37,66) | 20.50 (5.180) | 20.74 (5.491)
  Week 30: Emotional Well-Being (n=37,66) | 16.37 (4.164) | 17.23 (4.675)
  Week 30: Functional Well-Being (n=37,66) | 17.92 (5.082) | 17.93 (5.510)
  Week 30: FACT-L Subscale Score (n=37,66) | 25.90 (3.484) | 25.86 (4.817)
  Week 30: Lung Cancer Subscale Score (n=37,66) | 20.66 (3.073) | 20.61 (4.393)
  Week 30: Total FACT-G Score (n=37,66) | 76.54 (11.915) | 77.66 (15.078)
  Week 30: Trial Outcome Index (n=37,66) | 60.32 (9.753) | 60.30 (11.876)
  Week 30: Total FACT-L Score (n=37,66) | 102.44 (14.063) | 103.52 (18.367)
  Week 36: Physical Well-Being (n=25,47) | 21.60 (3.317) | 22.26 (4.480)
  Week 36: Social Well-Being (n=25,47) | 20.02 (5.769) | 20.15 (4.988)
  Week 36: Emotional Well-Being (n=25,47) | 17.31 (3.736) | 17.54 (4.540)
  Week 36: Fuctional Well-Being (n=25,47) | 16.06 (4.287) | 18.06 (5.720)
  Week 36: FACT-L Subscale Score (n=25,47) | 24.48 (4.089) | 25.83 (5.305)
  Week 36: Lung Cancer Subscale Score (n=25,47) | 19.36 (3.893) | 20.55 (4.463)
  Week 36: Total FACT-G Score (n=25,47) | 74.99 (11.066) | 78.02 (15.688)
  Week 36: Trial Outcome Index (n=25,47) | 57.02 (9.426) | 60.87 (11.963)
  Week 36: Total FACT-L Score (n=25,47) | 99.27 (13.672) | 103.86 (19.244)
  Week 42: Physical Well-Being (n=19,35) | 21.76 (3.592) | 22.19 (5.035)
  Week 42: Social Well-Being (n=19,35) | 18.45 (6.262) | 20.40 (5.234)
  Week 42: Emotional Well-Being (n=19,35) | 16.95 (4.089) | 17.43 (4.984)
  Week 42: Functional Well-Being (n=19,35) | 15.32 (3.902) | 18.57 (5.500)
  Week 42: FACT-L Subscale Score (n=19,35) | 24.63 (4.448) | 26.67 (5.357)
  Week 42: Lung Cancer Subscale Score (n=19,35) | 19.50 (4.092) | 21.21 (4.607)
  Week 42: FACT-G Score (n=19,35) | 72.74 (12.406) | 78.59 (16.316)
  Week 42: Trial Outcome Index (n=19,35) | 56.58 (9.562) | 61.97 (12.622)
  Week 42: FACT-L Score (n=19,35) | 97.11 (14.951) | 105.25 (20.385)
  Week 48: Physical Well-Being (n=13,29) | 21.38 (4.154) | 23.23 (4.016)
  Week 48: Social Well-Being (n=13,29) | 17.23 (7.567) | 20.24 (5.569)
  Week 48: Emotional Well-Being (n=13,29) | 18.69 (3.011) | 17.59 (4.903)
  Week 48: Functional Well-Being (n=13,29) | 14.15 (2.672) | 18.48 (4.501)
  Week 48: FACT-L Subscale Score (n=12,29) | 23.35 (3.647) | 26.80 (5.591)
  Week 48: Lung Cancer Subscale Score (n=12,29) | 18.75 (3.646) | 21.21 (4.967)
  Week 48: FACT-G Score (n=12,29) | 71.46 (12.069) | 79.53 (14.672)
  Week 48: Trial Outcome Index (n=12,29) | 54.58 (9.140) | 62.92 (11.105)
  Week 48: FACT-L Score (n=12,29) | 96.19 (14.394) | 106.33 (18.701)
  Week 60: Physical Well-Being (n=9,17) | 22.67 (4.664) | 23.65 (4.212)
  Week 60: Social Well-Being (n=9,17) | 17.78 (6.405) | 21.31 (6.530)
  Week 60: Emotional Well-Being (n=9,17) | 16.78 (3.232) | 19.12 (3.638)
  Week 60: Functional Well-Being (n=9,17) | 15.11 (3.408) | 18.65 (6.828)
  Week 60: FACT-L Subscale Score (n=9,17) | 23.43 (5.010) | 25.99 (6.844)
  Week 60: Lung Cancer Subscale Score (n=9,17) | 17.89 (3.919) | 20.47 (5.959)
  Week 60: Total FACT-G Score (n=9,17) | 72.34 (11.607) | 82.73 (17.803)
  Week 60: Trial Outcome Index (n=9,17) | 55.67 (9.695) | 62.76 (14.316)
  Week 60: Total FACT-L Score (n=9,17) | 95.77 (15.703) | 108.71 (23.069)
  Week 72: Physical Well-Being (n=6,8) | 22.17 (4.997) | 23.25 (4.097)
  Week 72: Social Well-Being (n=6,8) | 19.00 (7.251) | 21.44 (5.852)
  Week 72: Emotional Well-Being (n=6,8) | 17.17 (2.401) | 18.25 (5.007)
  Week 72: Functional Well-Being (n=6,8) | 15.22 (4.457) | 16.50 (5.855)
  Week 72: FACT-L Subscale Score (n=6,8) | 21.23 (5.154) | 26.48 (6.185)
  Week 72: Lung Cancer Subscale Score (n=6,8) | 17.17 (4.021) | 21.40 (5.724)
  Week 72: Total FACT-G Score (n=6,8) | 73.67 (14.820) | 79.44 (16.176)
  Week 72: Trial Outcome Index (n=6,8) | 54.67 (11.911) | 61.15 (14.343)
  Week 72: Total FACT-L Score (n=6,8) | 94.90 (18.833) | 105.92 (21.282)
  Week 84: Physical Well-Being (n=1,0) | 20.00 (NA) — Standard deviation (SD) not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants analyzed
  Week 84: Social Well-Being (n=1,0) | 14.00 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants analyzed
  Week 84: Emotional Well-Being (n=1,0) | 13.00 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants analyzed
  Week 84: Functional Well-Being (n=1,0) | 18.00 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants analyzed
  Week 84: FACT-L Subscale Score (n=1,0) | 17.00 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants analyzed
  Week 84: Lung Cancer Subscale Score (n=1,0) | 13.00 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants analyzed
  Week 84: Total FACT-G Score (n=1,0) | 65.00 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants analyzed
  Week 84: Trial Outcome Index (n=1,0) | 51.00 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants analyzed
  Week 84: Total FACT-L Score (n=1,0) | 82.00 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants analyzed
  Off Trtmt: Physical Well-Being (n=265,215) | 19.57 (5.668) | 18.50 (5.534)
  Off Trtmt: Social Well-Being (n=263,216) | 20.01 (5.380) | 20.68 (5.265)
  Off Trtmt: Emotional Well-Being (n=265,216) | 14.76 (5.157) | 15.11 (5.183)
  Off Trtmt: Functional Well-Being (n=265,216) | 14.90 (5.893) | 14.58 (5.934)
  Off Trtmt: FACT-L Subscale Score (n=264,214) | 22.80 (5.268) | 22.88 (4.911)
  Off Trtmt: Lung Cancer Subscale Score (n=264,214) | 18.06 (4.629) | 18.16 (4.383)
  Off Trtmt:Total FACT-G Score (n=261,214) | 69.29 (15.730) | 68.94 (15.669)
  Off Trtmt:Trial Outcome Index (n=263,213) | 52.61 (13.475) | 51.34 (12.974)
  Off Trtmt:Total FACT-L Score (n=260,212) | 92.14 (19.324) | 91.89 (18.738)

36. Secondary Outcome: Change From BL in FACT-L Scores (Data Cutoff 17 May 2008)
Description: as for outcome 35
Time Frame: as for outcome 2
Population: FAS; n=number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Number analyzed (Participants) | 274 | 303
score on a scale
  Week 6: Physical Well-Being (n=274,303) | 0.22 (4.235) | -0.47 (4.729)
  Week 6: Social Well-Being (n=274,303) | -0.24 (4.901) | 0.23 (4.202)
  Week 6: Emotional Well-Being (n=274,302) | -0.41 (3.801) | 0.29 (3.916)
  Week 6: Functional Well-Being (n=275,302) | 0.24 (4.819) | -0.09 (4.711)
  Week 6: FACT-L Subscale Score (n=275,298) | -0.06 (4.899) | 0.24 (4.623)
  Week 6: Lung Cancer Subscale Score (n=275,298) | -0.32 (4.148) | -0.03 (4.160)
  Week 6: Total FACT-G Score (n=273,299) | -0.20 (12.256) | 0.01 (11.453)
  Week 6: Trial Outcome Index (n=274,296) | 0.16 (10.276) | -0.73 (10.201)
  Week 6: Total FACT-L Score (n=273,294) | -0.20 (15.133) | 0.14 (14.155)
  Week 12: Physical Well-Being (n=144,193) | 1.00 (4.036) | -0.14 (4.908)
  Week 12: Social Well-Being (n=143,194) | -0.43 (4.918) | -0.43 (5.566)
  Week 12: Emotional Well-Being (n=144,194) | 0.25 (3.728) | 0.20 (4.115)
  Week 12: Functional Well-Being (n=144,196) | 1.00 (4.707) | -0.38 (4.806)
  Week 12: FACT-L Subscale Score (n=144,196) | 0.88 (4.501) | -0.06 (4.570)
  Week 12: Lung Cancer Subscale Score (n=144,196) | 0.19 (3.666) | -0.48 (4.004)
  Week 12: Total FACT-G Score (n=144,191) | 1.83 (11.637) | -0.84 (12.145)
  Week 12: Trial Outcome Index (n=144,193) | 2.20 (9.362) | -1.04 (10.051)
  Week 12: Total FACT-L Score (n=144,191) | 2.72 (14.226) | -0.90 (14.536)
  Week 18: Physical Well-Being (n=86,143) | 1.31 (4.798) | 0.40 (4.890)
  Week 18: Social Well-Being (n=86,143) | -0.01 (4.454) | -0.51 (5.894)
  Week 18: Emotional Well-Being (n=86,143) | 0.59 (3.984) | 0.60 (3.723)
  Week 18: Functional Well-Being (n=86,143) | 1.06 (4.353) | 0.18 (4.903)
  Week 18: FACT-L Subscale Score (n=86,143) | 1.48 (4.171) | 0.27 (4.587)
  Week 18: Lung Cancer Subscale Score (n=86,143) | 0.49 (3.550) | -0.26 (4.125)
  Week 18: Total FACT-G Score (n=86,143) | 2.95 (12.047) | 0.68 (12.668)
  Week 18: Trial Outcome Index (n=86,143) | 2.86 (9.638) | 0.32 (10.350)
  Week 18: Total FACT-L Score (n=86,143) | 4.43 (14.523) | 0.95 (15.386)
  Week 24: Physical Well-Being (n=59,101) | 1.29 (4.358) | 0.16 (4.881)
  Week 24: Social Well-Being (n=59,101) | -0.25 (4.804) | 0.04 (6.092)
  Week 24: Emotional Well-Being (n=59,100) | 0.21 (5.118) | -0.05 (4.169)
  Week 24: Functional Well-Being (n=59,100) | 1.64 (4.550) | 0.42 (4.373)
  Week 24: FACT-L Subscale Score (n=59,101) | 1.45 (5.018) | 0.50 (5.048)
  Week 24: Lung Cancer Subscale Score (n=59,101) | 0.48 (4.051) | -0.12 (4.321)
  Week 24: Total FACT-G Score (n=59,99) | 2.89 (13.739) | 0.52 (12.753)
  Week 24: Trial Outcome Index (n=59,100) | 3.42 (9.606) | 0.43 (10.348)
  Week 24: Total FACT-L Score (n=59,99) | 4.34 (16.354) | 1.10 (15.954)
  Week 30: Physical Well-Being (n=37,66) | 1.61 (4.205) | 0.49 (5.129)
  Week 30: Social Well-Being (n=37,66) | 0.00 (5.510) | -0.19 (6.676)
  Week 30: Emotional Well-Being (n=37,66) | -0.07 (4.902) | 0.74 (4.775)
  Week 30: Functional Well-Being (n=37,66) | 2.17 (5.028) | 0.83 (5.243)
  Week 30: FACT-L Subscale Score (n=37,66) | 1.79 (4.616) | 0.99 (4.863)
  Week 30: Lung Cancer Subscale Score (n=37,66) | 0.69 (3.818) | 0.38 (4.454)
  Week 30: Total FACT-G Score (n=37,66) | 3.71 (13.827) | 1.88 (14.268)
  Week 30: Trial Outcome Index (n=37,66) | 4.47 (9.551) | 1.70 (11.108)
  Week 30: Total FACT-L Score (n=37,66) | 5.50 (15.828) | 2.86 (16.864)
  Week 36: Physical Well-Being (n=25,47) | 2.21 (4.791) | 0.77 (5.093)
  Week 36: Social Well-Being (n=25,47) | -0.36 (5.659) | -0.16 (7.053)
  Week 36: Emotional Well-Being (n=25,47) | 0.86 (4.892) | 0.65 (3.717)
  Week 36: Functional Well-Being (n=25,47) | 1.31 (5.551) | 1.10 (5.280)
  Week 36: FACT-L Subscale Score (n=25,47) | 0.67 (4.864) | 0.43 (5.459)
  Week 36: Lung Cancer Subscale Score (n=25,47) | -0.10 (3.963) | -0.06 (4.535)
  Week 36: Total FACT-G Score (n=25,47) | 4.02 (14.439) | 2.37 (13.991)
  Week 36: Trial Outcome Index (n=25,47) | 3.42 (11.186) | 1.82 (10.443)
  Week 36: Total Fact-L Score (n=25,47) | 4.68 (17.636) | 2.79 (16.662)
  Week 42: Physical Well-Being (n=19,35) | 1.82 (3.936) | 0.27 (5.835)
  Week 42: Social Well-Being (n=19,35) | -1.14 (6.006) | 0.28 (7.784)
  Week 42: Emotional Well-Being (n=19,35) | -0.11 (3.573) | 0.59 (3.741)
  Week 42: Functional Well-Being (n=19,35) | 0.05 (3.582) | 0.65 (5.580)
  Week 42: FACT-L Subscale Score (n=19,35) | 1.40 (4.321) | 0.87 (4.974)
  Week 42: Lung Cancer Subscale Score (n=19,35) | 0.42 (2.858) | 0.51 (4.301)
  Week 42: FACT-G Score (n=19,35) | 0.62 (10.871) | 1.80 (15.245)
  Week 42: Trial Outcome Index (n=19,35) | 2.29 (7.037) | 1.44 (12.405)
  Week 42: FACT-L Score (n=19,35) | 2.03 (12.466) | 2.67 (18.499)
  Week 48: Physical Well-Being (n=13,29) | 0.46 (3.497) | 1.37 (6.388)
  Week 48: Social Well-Being (n=13,29) | -1.96 (7.987) | -0.68 (6.851)
  Week 48: Emotional Well-Being (n=13,29) | -0.08 (3.095) | 0.41 (4.166)
  Week 48: Functional Well-Being (n=13,29) | -2.00 (3.894) | 0.55 (5.448)
  Week 48: FACT-L Subscale Score (n=12,29) | 0.03 (4.445) | 0.82 (5.967)
  Week 48: Lung Cancer Subscale Score (n=12,29) | -0.79 (3.100) | 0.34 (5.150)
  Week 48: Total FACT-G Score (n=13,29) | -3.57 (12.233) | 1.64 (14.463)
  Week 48: Trial Outcome Index (n=12,29) | -1.79 (7.570) | 2.26 (13.247)
  Week 48: Total FACT-L Score (n=12,29) | -1.60 (11.354) | 2.46 (18.177)
  Week 60: Physical Well-Being (n=9,17) | 1.89 (5.383) | 1.82 (6.307)
  Week 60: Social Well-Being (n=9,17) | -0.57 (7.368) | 0.06 (9.116)
  Week 60: Emotional Well-Being (n=9,17) | -1.56 (2.789) | 0.28 (4.478)
  Week 60: Functional Well-Being (n=9,17) | -0.56 (3.877) | -0.53 (7.434)
  Week 60: FACT-L Subscale Score (n=9,17) | 1.61 (5.882) | 0.43 (6.275)
  Week 60: Lung Cancer Subscale Score (n=9,17) | -0.22 (4.438) | 0.47 (5.535)
  Week 60: Total FACT-G Score (n=9,17) | -0.79 (12.270) | 1.64 (17.542)
  Week 60: Trial Outcome Index (n=9,17) | 1.11 (11.044) | 1.76 (14.316)
  Week 60: Total FACT-L Score (n=9,17) | 0.82 (15.700) | 2.07 (22.086)
  Week 72: Physical Well-Being (n=6,8) | 1.33 (6.318) | 2.63 (7.130)
  Week 72: Social Well-Being (n=6,8) | 0.31 (6.723) | 0.30 (3.733)
  Week 72: Emotional Well-Being (n=6,8) | -1.50 (3.619) | -0.13 (4.853)
  Week 72: Functional Well-Being (n=6,8) | -1.67 (5.354) | -1.13 (5.384)
  Week 72: FACT-L Subscale Score (n=6,8) | -0.50 (7.396) | 1.03 (4.818)
  Week 72: Lung Cancer Subscale Score (n=6,8) | -1.17 (5.193) | 1.78 (4.141)
  Week 72: Total FACT-G Score (n=6,8) | -1.53 (11.929) | 1.67 (14.651)
  Week 72: Trial Outcome Index (n=6,8) | -1.50 (13.097) | 3.28 (13.738)
  Week 72: Total FACT-L Score (n=6,8) | -2.03 (16.140) | 2.70 (17.579)
  Week 84: Physical Well-Being (n=1,0) | 1.33 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants were analyzed
  Week 84: Social Well-Being (n=1,0) | -2.00 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants were analyzed
  Week 84: Emotional Well-Being (n=1,0) | -3.00 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants were analyzed
  Week 84: Functional Well-Being (n=1,0) | -1.00 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants were analyzed
  Week 84: FACT-L Subscale Score (n=1,0) | 6.0 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants were analyzed
  Week 84: Lung Cancer Subscale Score (n=1,0) | 2.0 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants were analyzed
  Week 84: Total FACT-G Score (n=1,0) | -4.67 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants were analyzed
  Week 84: Trial Outcome Index (n=1,0) | 2.33 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants were analyzed
  Week 84: Total FACT-L Score (n=1,0) | 1.33 (NA) — SD not calculated as only 1 participant was analyzed. | NA (NA) — Zero participants were analyzed
  Off Trtmt: Physical Well-Being (n=264,214) | -1.07 (4.750) | -2.19 (5.506)
  Off Trtmt: Social Well-Being (n=263,216) | -0.66 (4.973) | 0.09 (4.824)
  Off Trtmt: Emotional Well-Being (n=264,216) | -2.04 (4.225) | -1.56 (4.745)
  Off Trtmt: Functional Well-Being (n=264,216) | -1.20 (5.170) | -1.98 (5.355)
  Off Trtmt: FACT-L Subscale Score (n=263,212) | -1.27 (4.458) | -1.32 (4.708)
  Off Trtmt: Lung Cancer Subscale Score (n=263,212) | -1.74 (3.882) | -1.78 (4.199)
  Off Trtmt: Total FACT-G Score (n=260,213) | -4.91 (12.576) | -5.71 (13.588)
  Off Trtmt: Trial Outcome Index (n=261,210) | -4.03 (10.658) | -6.05 (11.785)
  Off Trtmt: Total FACT-L Score (n=258,209) | -6.26 (15.146) | -7.10 (16.194)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from Day 1 (after randomization) through the end of study, up to 27 months. Serious adverse events (SAEs) were recorded from Day 1 (after randomization) through the second data cut-off, up to 71 months.
Description: All participants who received at least 1 dose of investigational treatment and had at least 1 safety follow-up, whether prematurely withdrawn or not, were included in the safety analysis.
Arm/Group | Placebo | Erlotinib, 150 mg/Day
Serious Adverse Events (participants affected / at risk) | 34/445 | 49/433
Other Adverse Events (participants affected / at risk) | 152/445 | 283/433
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=445) | Erlotinib, 150 mg/Day (N=433)
Pneumonia (Infections and infestations) | 4 | 7
Bronchitis (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Catheter sepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2
Empyema (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1
Nocardiosis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Colitis (Infections and infestations) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Vomiting (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Urogenital haemorrhage (Renal and urinary disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Drowning (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Aortic aneurysm (Cardiac disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 1
Arterial thrombosis (Vascular disorders) | 1 | 0
Arteritis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Iliac artery thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=445) | Erlotinib, 150 mg/Day (N=433)
Rash (Skin and subcutaneous tissue disorders) | 26 | 211
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 32
Acne (Skin and subcutaneous tissue disorders) | 0 | 27
Diarrhoea (Gastrointestinal disorders) | 20 | 87
Nausea (Gastrointestinal disorders) | 27 | 33
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 36
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 37 | 33
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 21 | 22
Fatigue (General disorders) | 26 | 39
Chest pain (General disorders) | 28 | 14
Anorexia (Metabolism and nutrition disorders) | 22 | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.